CLINICAL TRIAL: NCT01835496
Title: The Pharmacokinetic Profile of a Single Dose of Ferriprox® in Patients With Sickle Cell Disease
Brief Title: Absorption, Metabolism, and Excretion of a Single Dose of Ferriprox® in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: LA41-0412
Record Dates: First submitted 2013-04-11; First posted 2013-04-19 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2013-04

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; iron overload; pharmacokinetics; Ferriprox; deferiprone
MeSH Terms: conditions — Anemia, Sickle Cell; Iron Overload | interventions — Single Person; Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferriprox (No Intervention): single 1500 mg dose of Ferriprox
  Interventions: Drug: single 1500 mg dose of Ferriprox

INTERVENTIONS:
Drug: single 1500 mg dose of Ferriprox — A single dose of 1500mg of Ferriprox (three 500mg tablets) administered under fasting conditions
  Other Names: deferiprone

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics of deferiprone and its 3-O-glucuronide metabolite following administration of a single 1500 mg dose of Ferriprox in patients with sickle cell disease.

DETAILED DESCRIPTION:
This is a single-arm, single-dose study of Ferriprox in patients with sickle cell disease. Patients found to be eligible will visit the clinic the day before receiving the drug, in order to reconfirm eligibility and to undergo baseline assessments, and will receive a single dose of 1500 mg Ferriprox under fasting conditions. Blood and urine samples for pharmacokinetic assessment will be collected over a 10-hour period. Standard safety assessments will be performed throughout the study, and patients will return for a safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-45 years of age (inclusive)
2. Diagnosis of sickle cell disease, confirmed by Hb electrophoresis
3. Body weight ≥ 50 kg
4. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m^2
5. Absolute neutrophil count (ANC) of >1.5 x 10^9/L
6. Women of childbearing potential must agree to either be sexually inactive or use an acceptable method of birth control for 14 days prior to dosing and for 30 days afterwards
7. A fertile heterosexual male must agree that he or his partner will use an effective method of contraception for 14 days prior to dosing and for 30 days afterwards

Exclusion Criteria:

1. History or presence of hypersensitivity or idiosyncratic reaction to Ferriprox
2. Use of Ferriprox within the past 3 months
3. History of malignancy
4. Evidence of abnormal liver function (serum Alanine Transaminase (ALT)level > 5 times upper limit of normal or creatinine levels >2 times upper limit of normal)
5. A serious, unstable illness, as judged by the Investigator, within the past 3 months before screening visit including but not limited to hepatic, renal, gastro-enterologic, respiratory, cardiovascular, endocrinologic, neurologic or immunologic disease
6. Hemodialysis during the week prior to dosing or planned for the day of dosing
7. Known difficulty in providing blood samples
8. Disorders or surgery of the gastrointestinal tract that may interfere with drug absorption or may otherwise influence the Pharmacokinetic (PK) results (e.g., resection of the small or large intestine, febrile conditions, chronic diarrhea, chronic vomiting, endocrine disease, severe infections, acute inflammations, etc.)
9. Clinically significant abnormalities on 12-lead ECG (e.g., QT interval corrected using Fridericia's formula (QTcF) ≥ 430 ms in males or ≥ 450 ms in females)
10. Use of tobacco/nicotine-containing products for at least 3 months prior to study drug administration
11. Use of any drugs within the past 14 days that are metabolized by the Uridine diphosphate glucosyltransferase enzyme (UGT1A6) and hence could affect the PK of Ferriprox
12. Treatment with an investigational drug within the past 30 days or 5 half-lives of that drug (whichever is longer) prior to study drug administration
13. Pregnant or nursing female

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Soulieres, MD, Principal Investigator — CHUM - Hôpital Notre-Dame
Locations (1):
- CHUM-Hôpital Notre-Dame, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Soulieres D, Mercier-Ross J, Fradette C, Rozova A, Tsang YC, Tricta F. The pharmacokinetic and safety profile of single-dose deferiprone in subjects with sickle cell disease. Ann Hematol. 2022 Mar;101(3):533-539. doi: 10.1007/s00277-021-04728-0. Epub 2022 Jan 4. PMID 34981144

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferriprox: A single dose of 1500 mg of Ferriprox (three 500 mg tablets) administered under fasting conditions
Period: Overall Study
Arm/Group | Ferriprox
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  Canada | 8

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: Cmax (maximum measured serum concentration) was assessed over a 10-hour interval for deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained pre-dose and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, and 10 hours post-dose.
Time Frame: 10-hour interval
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
μg/mL
  Cmax for serum deferiprone | 17.56 (5.76)
  Cmax for serum deferiprone 3-O-glucuronide | 32.95 (11.85)

2. Secondary Outcome: Frequency of Adverse Events
Time Frame: From Day 1 (Dosing) to Day 7 plus/minus 3 days (Follow-up)
Measure: Number; unit: participants
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
participants | 2

3. Secondary Outcome: Frequency of Serious Adverse Events
Time Frame: From Day 1 (Dosing) to Day 30 post-dose
Measure: Number; unit: participants
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
participants | 0

4. Primary Outcome: Tmax for Deferiprone and Deferiprone 3-O-glucuronide
Description: Tmax (time to the maximum measured serum concentration) was assessed over a 10-hour interval for deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained pre-dose and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, and 10 hours post-dose.
  The results of the Tmax parameter are reported as the median and range (other parameters are reported as mean and standard deviation).
Time Frame: 10-hour interval
Measure: Median (Full Range); unit: hr
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
hr
  Tmax for serum seferiprone | 1.000 [0.50 to 2.50]
  Tmax for serum deferiprone 3-O-glucuronide | 2.750 [1.33 to 3.00]

5. Primary Outcome: AUC0-∞ for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: AUC0-∞ (area under the curve, zero to infinity) was assessed over a 10-hour interval for deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained pre-dose and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, and 10 hours post-dose.
Time Frame: 10-hour interval
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
µg*hr/mL
  AUC0-∞ for serum deferiprone | 43.37 (5.39)
  AUC0-∞ for serum deferiprone 3-O-glucuronide | 142.7 (47.02)

6. Primary Outcome: T1/2 for Serum Deferiprone and Deferiprone 3-O-glucuronide
Description: T1/2 (apparent terminal elimination half-life) was assessed over a 10-hour interval for deferiprone and its 3-O-glucuronide metabolite. Blood samples were obtained pre-dose and at 0.25, 0.50, 0.75, 1, 1.33, 1.66, 2, 2.5, 3, 4, 6, 8, and 10 hours post-dose.
Time Frame: 10-hour interval
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Ferriprox
Number analyzed (Participants) | 8
hr
  T1/2 for serum deferiprone | 1.458 (0.207)
  T1/2 for serum deferiprone 3-O-glucuronide | 1.575 (0.217)

ADVERSE EVENTS:
Time Frame: From the time of dosing to 7 ±3 days post-dose
Arm/Group | Ferriprox
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferriprox (N=8)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All unpublished information given to the PI by ApoPharma shall not be published or disclosed to a third party without the prior written consent of ApoPharma.

The data generated by this study are considered confidential information and the property of ApoPharma. This confidential information may be published only in collaboration with participating personnel from ApoPharma or upon ApoPharma written consent to publish the article.